CLINICAL TRIAL: NCT07176572
Title: Comparison of Analgesic Efficacy of Transcutaneous Electrical Nerve Stimulation and Dexketoprofen Trometamol in Patients Presenting to the Emergency Department With Renal Colic: A Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Transcutaneous Electrical Nerve Stimulation and Dexketoprofen in Renal Colic
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Professor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RK-TENSE-2025-AEAH
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Renal Colic
Keywords: Transcutaneous electrical nerve stimulation; emergency medicine; Dexketoprofen Trometamol
MeSH Terms: conditions — Renal Colic | interventions — Transcutaneous Electric Nerve Stimulation; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Transcutaneous electrical nerve stimulation (TENS) (Experimental): Patients receiving the real transcutaneous electrical nerve stimulation (TENS) with 100 hertz, pulse width 200 microseconds, voltage 2 milliampere
  Interventions: Device: TENS
- dexketoprofen trometamol (Active Comparator): 50 mg dexketoprofen trometamol
  Interventions: Drug: Dexketoprofen Trometamol

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation (TENS) treatment will be activated + NS IV Infusion 100 ml
  Other Names: Comfort plus TENS device
  Arms: Real Transcutaneous electrical nerve stimulation (TENS)
Drug: Dexketoprofen Trometamol — 50 mg dexketoprofen trometamol in 100 ml normal saline solution + Transcutaneous electrical nerve stimulation treatment will not be activated.
  Other Names: Ketavel (dexketoprofen trometamol)
  Arms: dexketoprofen trometamol

SUMMARY:
The aim of this study was to compare the analgesic efficacy of transcutaneous electrical nerve stimulation (TENS) and dexketoprofen trometamol in patients presenting to the emergency department due to renal colic.

DETAILED DESCRIPTION:
Renal colic is a common presenting complaint to the emergency department and is an intensely painful condition. Parenteral opioids, non-steroidal anti-inflammatory drugs (NSAIDs) and paracetamol are commonly used to relieve the pain of renal colic. Dexketoprofen trometamol is a non-steroidal anti-inflammatory drug that is frequently used in the management of acute pain. Common and known side effects of nonsteroidal anti-inflammatory drugs include gastrointestinal system problems and allergic reactions. Transcutaneous electrical nerve stimulation is a non-invasive, non-pharmacological and low-risk treatment method. This study aimed to compare the analgesic efficacy of Transcutaneous electrical nerve stimulation and dexketoprofen trometamol in patients presenting to the emergency department with renal colic.

Study Design and Setting: A prospective, randomized, double-blind, single-center, clinical trial will be conducted in emergency department of a tertiary care university hospital.

Statistical Analysis:

Categorical variables will be presented as numbers and percentages. The Kolmogorov-Smirnov test will be used to evaluate the normality of the distribution of continuous variables. Continuous variables with a non-normal distribution will be expressed as the median and interquartile range (IQR), and those with a normal distribution will be expressed as the mean and standard deviation (SD). The Mann-Whitney U test will be used to analyse non-normally distributed variables to evaluate the differences in visual analog scale scores between the two groups; the Student's t-test will be used for normally distributed variables.

The sample size was calculated using the G*Power 3.1.9.2 programme. According to the data obtained from the study of renal colic therapy with TENS, a difference of 18.4 mm in visual analogue scale score between the two groups with a standard deviation of 6 mm was assumed. It was calculated that 64 patients were required for each group with a two-sided critical value of α = 0.05, 95% power and an effect size of 0.5.

ELIGIBILITY:
Inclusion Criteria:

- Aged 18 years or over with a definite diagnosis of renal colic

Exclusion Criteria:

* Patients who refuse to participate in the study
* Pregnant women
* Breastfeeding women
* Haemodynamically unstable
* Evidence of peritoneal inflammation
* Patients who were taking analgesics at the time of initial presentation
* Unconsciousness or inability to communicate
* Contraindications to applying TENS or using the drug in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the intensity of pain | 15 minutes and 30 minutes after the administration of the study interventions
  Pain intense will be measured by 100 mm visual analog scale (Zero; no pain and 100 mm; the worst pain) after 15th and 30th minutes later the administration of the study interventions

SECONDARY OUTCOMES:
Adverse events | 30 minutes after
  30 minutes after the administration of the study interventions
need to rescue medication | 30 minutes after
  30 minutes after the administration of the study interventions

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Prof.Dr., Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Medical Faculty, Adıyaman, Turkey (Türkiye)

REFERENCES:
- [Background] Gulacti U, Algin A, Turgut K, Yavuz E, Aydin I, Buyukaslan H, Lok U, Arslan E, Gonel A. Transcutaneous Electrical Nerve Stimulation (TENS) for the Treatment of Renal Colic in the ED: A Randomized, Double-Blind, Placebo-Controlled Trial. Am J Emerg Med. 2022 Jun;56:127-132. doi: 10.1016/j.ajem.2022.02.044. Epub 2022 Mar 29. PMID 35397352
- [Background] Al B, Sunar MM, Zengin S, Sabak M, Bogan M, Can B, Kul S, Murat Oktay M, Eren SH. Comparison of IV dexketoprofen trometamol, fentanyl, and paracetamol in the treatment of renal colic in the ED: A randomized controlled trial. Am J Emerg Med. 2018 Apr;36(4):571-576. doi: 10.1016/j.ajem.2017.09.019. Epub 2017 Sep 14. PMID 29029797
- [Background] Hanna M, Moon JY. A review of dexketoprofen trometamol in acute pain. Curr Med Res Opin. 2019 Feb;35(2):189-202. doi: 10.1080/03007995.2018.1457016. Epub 2018 Apr 24. PMID 29569951